CLINICAL TRIAL: NCT04312737
Title: European VALidation of HUman Papillomavirus Assays and Collection DEvices for HPV Testing on Self-samples and Urine Samples
Brief Title: Evaluation of in Vitro Devices on Self-collected Vaginal Swab and Urine Sample for Testing of Human Papilloma Virus
Acronym: EU-VALHUDES
Status: Completed | Type: Observational
Sponsor: Hiantis Srl (Industry)
Collaborators: Genefirst LTD (Unknown); Sciensano (Other Government)
Responsible Party: Sponsor
Other Study IDs: WP6-HPVONC; GA-806551 (Other Grant/Funding Number: Horizon 2020 SME Instrument Project)
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; Neoplasm Cervix; Carcinoma in Situ; Carcinoma Cervix Uterine; Neoplasms; Neoplasms by Histologic Type
Keywords: self-sampling; HPV testing; Diagnostic Test Accuracy; Cervical Intraepithelial Neoplasia; Urine; Cervical Cancer Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Carcinoma in Situ; Neoplasms; Neoplasms by Histologic Type; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Urine, vaginal and cervical samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Self-Collecting Devices — FLOQSwab (Copan) Colli-Pee (Novosanis)
Diagnostic Test: In Vitro Diagnostic Assays — Papilloplex (GeneFirst) HPV Oncopredict DNA (Hiantis) HPV Oncopredict RNA (GeneFirst)

SUMMARY:
The European VALHUDES study is a Clinical Performance /Diagnostic Test Accuracy Study that aims to evaluate whether HPV testing with new assays performed on self-samples, collected by means of a vaginal and a urine collection device is as accurate to detect cervical pre-cancer as on cliniciantaken cervical samples.

DETAILED DESCRIPTION:
Women accessing the Colposcopy Centres for a colposcopy examination and fulfilling the selection criteria will be asked, after written informed consent, to self-collect a first-void urine (with the Colli-Pee device) and a vaginal sample (with the FLOQSwab device), prior to undergoing colposcopy. Just before colposcopic examination, a clinician will also take a cervical sample (with a Cervex-Brush using the same procedure normally adopted for cervical cytology and/or HPV testing. During colposcopy, a colposcopy-targeted biopsy may be taken if appropriate. When according to colposcopy and biopsy results, an excisional treatment of a cervical precancer lesion is needed, the histology of the excised tissue will complete the end point of the study. The colposcopy and histological findings will be used as the gold standard if biopsies are taken.

In case of normal satisfactory colposcopic findings without biopsy taking, colposcopy will provide the study outcome.

Three new PCR-based HPV 'in vitro diagnostic devices' (Papilloplex, HPV Oncopredict RNA, HPV Oncopredict DNA) developed as part of the SME Instrument Project 'HPV OncoPredict (GA-806551)' will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women referred to colposcopy evaluation for any reason [i.e. previous history of abnormal cervical screen test results (cytology, HPV test), previous abnormal colposcopy]
* Ability to understand and sign the informed consent
* Informed consent given

Exclusion Criteria:

* Age < 25 or > 65 years
* Past history of hysterectomy
* Women with known pregnancy
* Pregnancy within last 3 months
* Vulnerable patient: a patient who is or may be for any reason unable to take care of him or herself, or unable to protect him or herself against significant harm or exploitation
* Simultaneous involvement in any other research project

Ages: 25 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women referred to colposcopy evaluation for any reason [i.e. previous history of abnormal cervical screen test results (cytology, HPV test), previous abnormal colposcopy]
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Relative accuracy urine vs clinician-collected samples | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Relative sensitivity and specificity of each hrHPV DNA assay for detection of cervical intraepithelial neoplasia of grade II or worse (CIN2+) on urine vs on clinician-collected samples.
Relative accuracy self-collected vaginal vs clinician-collected samples | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Relative sensitivity and specificity of each hrHPV DNA assay for detection of cervical intraepithelial neoplasia of grade II or worse (CIN2+) on self-collected vaginal vs on clinician-collected samples.

SECONDARY OUTCOMES:
Absolute accuracy for each sample type | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Absolute clinical sensitivity and specificity for finding underlying CIN2/3+ of the investigated hrHPV assays applied on each sample.
Absolute accuracy among hrHPV DNA-positive women | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Absolute clinical sensitivity and specificity using HPV OncoPredict RNA among women with hrHPV DNA-positive result on one of the self-samples.
Concordance of presence or absence of HPV genotypes between different sample types | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Concordance of presence of hrHPV and of HPV genotypes between urine, vaginal and clinician-collected samples.
Correlation viral load signals between different sample types | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Correlation of genotype-specific viral load signals between urine, vaginal and clinician-collected samples.
Concordance of presence or absence of internal control gene between different sample types | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Concordance of positivity for the human cellular control between urine, vaginal and clinician-collected samples.
Correlation internal control gene signals between different sample types | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Correlation of signals for the human internal control gene between urine, vaginal and clinician-collected samples.
Positivity rates human control gene | One day, with possible extension if excision biopsy is planned based on the coloposcopy/histology outcome of tissue specimens collected at the enrolment visit.
  Positivity rates for human cellular control in the different sample types.
Questionnaire for the acceptance of self-collection | One day, at the day of colposcopy
  Women's acceptance and preference regarding urine collection, vaginal self-sampling or collection by a clinician will be assessed through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Arbyn, Dr, Principal Investigator — Sciensano
Locations (6):
- The Coombe Women and Infants University Hospital, & Trinity College, Dublin, Ireland
- Italy (4):
  - Dipartimento di Chirurgia e Medicina - Università Milano-Bicocca, Monza, Monza Brianza
  - Spedali Civili di Brescia, Brescia
  - European Institute of Oncology, Milan
  - ATS-Sardegna Azienda Tutela Salute. ASSL Sassari, Sassari
- Scottish HPV Reference Laboratory, Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Result] Arbyn M, Peeters E, Benoy I, Vanden Broeck D, Bogers J, De Sutter P, Donders G, Tjalma W, Weyers S, Cuschieri K, Poljak M, Bonde J, Cocuzza C, Zhao FH, Van Keer S, Vorsters A. VALHUDES: A protocol for validation of human papillomavirus assays and collection devices for HPV testing on self-samples and urine samples. J Clin Virol. 2018 Oct;107:52-56. doi: 10.1016/j.jcv.2018.08.006. Epub 2018 Aug 22. PMID 30195193